CLINICAL TRIAL: NCT05030584
Title: A Double-blind, Randomized, Placebo-controlled Multicenter Study to Investigate Efficacy and Safety of Elinzanetant for the Treatment of Vasomotor Symptoms Over 52 Weeks in Postmenopausal Women
Brief Title: A Study to Learn More About How Well Elinzanetant Works and How Safe it is for the Treatment of Vasomotor Symptoms (Hot Flashes) That Are Caused by Hormonal Changes Over 52 Weeks in Women Who Have Been Through the Menopause
Acronym: OASIS-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21810; 2021-000059-38 (EudraCT Number)
Record Dates: First submitted 2021-08-27; First posted 2021-09-01 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Vasomotor Symptoms Associated With Menopause; Hot Flashes
Keywords: Menopause
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elinzanetant (BAY3427080) (Experimental): Participants will receive 120 mg elinzanetant orally once daily.
  Interventions: Drug: Elinzanetant (BAY3427080)
- Placebo (Placebo Comparator): Participants will receive matching placebo orally once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — 120 mg elinzanetant orally once daily
  Arms: Elinzanetant (BAY3427080)
Drug: Placebo — Matching placebo orally once daily.
  Arms: Placebo

SUMMARY:
Researchers are looking for a better way to treat women who have hot flashes after they have been through the menopause. Hot flashes are caused by the hormonal changes that happen when a woman's body has been through the menopause. Menopause is when women stop having a menstrual cycle, also called a period. During the menopause, the ovaries increasingly produce less sex hormones as a result of the natural ageing process and related hormonal adjustments. The decline in hormone production can lead to various symptoms which, in some cases, can have a very adverse effect on a menopausal woman's quality of life.

The study treatment, elinzanetant, was developed to treat symptoms caused by hormonal changes. It works by blocking a protein called neurokinin from sending signals to other parts of the body, which is thought to play a role in starting hot flashes. There are treatments for hot flashes in women who have been through the menopause, but may cause medical problems for some people.

In this study, the researchers will learn how well elinzanetant works compared to a placebo in women who have been through the menopause and have hot flashes. A placebo is a treatment that looks like a medicine but does not have any medicine in it. To compare these study treatments, the participants will record information about their hot flashes in an electronic diary. The researchers will study the number of hot flashes the participants have and how severe they are. They will study the results from before treatment and after 12 weeks of treatment.

The participants in this study will take two capsules of either elinzanetant or the placebo once a day. The participants will take the study treatments for 52 weeks.

During the study, the participants will visit their study site approximately 11 times and perform 2 visits by phone. Each participant will be in the study for approximately 62 weeks.

During the study, the participants will:

* record information about their hot flashes in an electronic diary
* answer questions about their symptoms

The doctors will:

* check the participants' health
* take blood samples
* ask the participants questions about what medicines they are taking and if they are having adverse events An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, defined as:

  1. at least 12 months of spontaneous amenorrhea prior to signing of informed consent, or
  2. at least 6 months of spontaneous amenorrhea prior to signing of informed consent with serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL and a serum estradiol concentration of < 30 pg/mL, or
  3. at least 6 months after hysterectomy at signing of informed consent with serum FSH levels > 40 mIU/mL and a serum estradiol concentration of < 30 pg/mL, or
  4. surgical bilateral oophorectomy with or without hysterectomy at least 6 weeks prior to signing of informed consent.
* Moderate to severe hot flash (HF) associated with the menopause and seeking treatment for this condition.
* Participant has completed Hot Flash Daily Diary (HFDD) for at least 11 days during the two weeks preceding baseline visit and is showing eligibility with respect to previous inclusion criterion during this time period.

Exclusion Criteria:

* Any clinically significant prior or ongoing history of arrhythmias, heart block and QT prolongation either determined through clinical history or on ECG evaluation.
* Any active ongoing condition that could cause difficulty in interpreting vasomotor symptoms (VMS) such as: infection that could cause pyrexia, pheochromocytoma, carcinoid syndrome.
* Current or history (except complete remission for 5 years or more) of any malignancy (except basal and squamous cell skin tumors). Women receiving adjuvant endocrine therapy (e.g. tamoxifen, aromatase inhibitors, GnRH analogues) cannot be enrolled in this study.
* Uncontrolled or treatment-resistant hypertension. Women with mild hypertension can be included in the study if they are medically cleared prior to study participation.
* Untreated hyperthyroidism or hypothyroidism.

  * Treated hyperthyroidism with no abnormal increase of thyroid function laboratory parameters and no relevant clinical signs for > 6 months before signing of informed consent is acceptable.
  * Treated hypothyroidism with normal thyroid function test results during screening and a stable (for ≥ 3 months before signing of informed consent) dose of replacement therapy is acceptable.
* Any unexplained post-menopausal uterine bleeding
* Clinically relevant abnormal findings on mammogram.
* Abnormal liver parameters.
* Disordered proliferative endometrium, endometrial hyperplasia, polyp, or endometrial cancer diagnosed based on endometrial biopsy during screening.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2024-02-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (86):
- United States (36):
  - Mobile ObGyn, P.C. | Mobile, AL, Mobile, Alabama
  - Mesa Obstetricians and Gynecologists | Research Department, Mesa, Arizona
  - National Institute of Clinical Research - Garden Grove, Garden Grove, California
  - Marvel Clinical Research | Huntington Beach, CA, Huntington Beach, California
  - Empire Clinical Research | Pomona, CA, Pomona, California
  - Coastal Connecticut Research | New London, CT, New London, Connecticut
  - IntimMedicine | Washington, DC, Washington D.C., District of Columbia
  - Boca Midwifery, Boca Raton, Florida
  - Helix Biomedics LLC | Boynton Beach, FL, Boynton Beach, Florida
  - UF Health Women's Specialists - Emerson, Jacksonville, Florida
  - Suncoast Clinical Research - Palm Harbor, Palm Harbor, Florida
  - Physician Care Clinical Research LLC | Sarasota, FL, Sarasota, Florida
  - Suncoast Clinical Research - New Port Richey, Trinity, Florida
  - Paramount Research Solutions | College Park Location, College Park, Georgia
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Southern Clinical Research, LLC, Zachary, Louisiana
  - Johns Hopkins Hospital - Gynecology and Obstetrics, Baltimore, Maryland
  - Boeson Research | Great Falls, MT, Great Falls, Montana
  - Boeson Research | Missoula, MT, Missoula, Montana
  - Affiliated Clinical Research, Inc. | Las Vegas, NV, Las Vegas, Nevada
  - AMR - Las Vegas, Las Vegas, Nevada
  - Elite Clinical Network (ECN) | Las Vegas Clinical Trials, LLC, North Las Vegas, Nevada
  - M3 Wake Research | Raleigh, NC, Raleigh, North Carolina
  - ClinOhio Research Services, LLC. | Columbus, OH, Columbus, Ohio
  - HWC Women's Research Center | Englewood, OH, Englewood, Ohio
  - Clinical Research Philadelphia | Philadelphia, PA, Philadelphia, Pennsylvania
  - Venus Gynecology, LLC | Myrtle Beach, SC, Myrtle Beach, South Carolina
  - Advances in Health, INC. | Houston, TX, Houston, Texas
  - UTHealth Womens Research Program | Memorial City, Houston, Texas
  - Elligo Health Research | Medical Colleagues of Texas, Hurst, Texas
  - Elligo Health Research | Protenium Clinical Research, Katy, Texas
  - Maximos Ob/Gyn, League City, Texas
  - Tidewater Clinical Research - Norfolk, Norfolk, Virginia
  - Eastern Virginia Medical School | OB/GYN Clinical Research Center, Norfolk, Virginia
  - Seattle Clinical Research Center, Seattle, Washington
- Belgium (5):
  - CHU Saint-Pierre/UMC Sint-Pieter, Bruxelles - Brussel
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liege | CHR Citadel - Department of Gyneacology and Obstetrics, Liège
  - Femicare vzw | Tienen, BE, Tienen
- Bulgaria (11):
  - Medical Centre Asklepii OOD | Dupnitsa, Bulgaria, Dupnitsa
  - Multiprofile Hospital for Active Treatment | Avis Medica - Obstetrics and Gynecology, Pleven
  - Multiprofile Hospital for Active Treatment Plovdiv | Obstetrics and Gynecology, Plovdiv
  - Spec.Hospital for obstetrics and gynecology Selena OOD, Plovdiv
  - Multiprofile Hospital for Active Treatment Samokov | Gynecology Department, Samokov
  - Specialized Hospital for Active Treatment of Oncological Diseases Sofia Region | Oncological Gynecology Department, Sofia
  - Multiprofile Hospital for Active Treatment for Women's Health Nadezhda | Department of Obstetrics and Gynecology, Sofia
  - Diagnostic-Consultative Center Alexandrovska | Sofia, Bulgaria, Sofia
  - Medical Center Panacea OOD | Sofia, Bulgaria, Sofia
  - Multiprofile Hospital for Active Treatment Niamed OOD | Department of Obstetrics and Gynecology, Stara Zagora
  - SBAGAL Dr. Dimitar Stamatov | Varna, Bulgaria, Varna
- Canada (8):
  - IWK Health Centre | Department of Obstetrics and Gynaecology, Halifax, Nova Scotia
  - Manna Research (Burlington North), Burlington, Ontario
  - Manna Research (Ottawa), Nepean, Ontario
  - Ottawa Hospital-Riverside Campus, Ottawa, Ontario
  - Viable Clinical Research | Mississauga, Canada, Scarborough Village, Ontario
  - Manna Research (Quebec), Lévis, Quebec
  - Manna Research (Montreal), Pointe-Claire, Quebec
  - Alpha Recherche Clinique | Lebourgneuf, Québec
- Denmark (3):
  - Sanos Clinic | Gandrup, Denmark, Gandrup
  - Sanos Clinic | Herlev, Denmark, Herlev
  - Sanos Clinic | Syddanmark, Vejle, Denmark, Vejle
- Finland (5):
  - HUS / Naistenklinikka, Helsinki
  - Pihlajalinna Lääkärikeskus Oy, Savo-Karjala, Joensuu
  - Mehilainen | Mehilainen Kuopio, Kuopio
  - Lääkärikeskus Gyneko, Gynaecological Medical Center | Oulu, Finland, Oulu
  - Terveystalo | Terveystalo Tampere Research Unit, Tampere
- Poland (6):
  - Gabinet Ginekologiczny Janusz Tomaszewski, Bialystok
  - CLINICAL MEDICAL RESEARCH Sp. z o. o., Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Badawcze Wspolczesnej Terapii, Warsaw
- Spain (7):
  - Hospital Universitario La Zarzuela - Ginecologia, Aravaca, Madrid
  - Hospital de la Santa Creu i Sant Pau | Gynecology Department, Barcelona
  - Instituto Palacios | Investigation Research Unit - Gynecology department, Madrid
  - Hospital Clinico San Carlos | Women´s Health Institute, Madrid
  - Hospital Universitario 12 de Octubre | Department of Obstetrics and Gynecology, Madrid
  - Virgen del Rocio University Hospital | Gynecology Unit, Seville
  - Hospital Clinico Universitario | Gynecology and Obstetrics Department, Valencia
- United Kingdom (5):
  - MAC Clinical Research | Lancashire - Clinical Research Centre, Blackpool
  - NHS Greater Glasgow and Clyde | Glasgow Royal Infirmary - Gynaecology, Glasgow
  - Liverpool Women's NHS Foundation Trust | Liverpool Women's Hospital - Gynaecology, Liverpool
  - Imperial College Healthcare NHS Trust| Queen Charlotte's and Chelsea Hospital - Gynaecology, London
  - MAC Clinical Research | Greater Manchester Early Phase - Clinical Research Centre, Manchester

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Panay N, Joffe H, Maki PM, Nappi RE, Pinkerton JV, Simon JA, Soares CN, Thurston RC, Francuski M, Caetano C, Genga K, Haberland C, Haseli Mashhadi N, Laapas K, Parke S, Seitz C, Schwarz J, Zuurman L. Elinzanetant for the Treatment of Vasomotor Symptoms Associated With Menopause: A Phase 3 Randomized Clinical Trial. JAMA Intern Med. 2025 Nov 1;185(11):1319-1327. doi: 10.1001/jamainternmed.2025.4421. PMID 40920404
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/21810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 75 study centers in North America and in several countries in Europe, between 27-Aug-2021 (first participant first visit) and 12-Feb-2024 (last participant last visit).
Pre-assignment Details: A total of 1524 patients were screened, of whom 628 were randomized.
Groups:
- Elinzanetant (BAY3427080): Participants received 120 mg elinzanetant orally once daily.
- Placebo: Participants received matching placebo orally once daily.
Period: Overall Study
Arm/Group | Elinzanetant (BAY3427080) | Placebo
Started | 313 | 315
Received Treatment | 312 | 315
Completed | 222 | 231
Not Completed | 91 | 84
Not completed — Adverse Event | 17 | 2
Not completed — Lack of Efficacy | 0 | 6
Not completed — Lost to Follow-up | 5 | 2
Not completed — Non-Compliance with Study Drug | 2 | 3
Not completed — Other reason | 4 | 3
Not completed — Physician Decision | 1 | 4
Not completed — Protocol Violation | 0 | 2
Not completed — Randomized by Mistake | 0 | 2
Not completed — Withdrawal by Subject | 21 | 28
Not completed — Technical Problems | 0 | 1
Not completed — Completed post-treatment/FU visits | 41 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elinzanetant (BAY3427080) | Placebo | Total
Number analyzed (Participants) | 313 | 315 | 628
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (4.7) | 54.9 (5.0) | 54.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 313 | 315 | 628
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 34 | 68
  Not Hispanic or Latino | 266 | 273 | 539
  Unknown or Not Reported | 13 | 8 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 51 | 44 | 95
  White | 240 | 253 | 493
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 19 | 15 | 34

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Frequency of Moderate to Severe Hot Flashes (HFs) From Baseline to Week 12 (Assessed by Hot Flash Daily Diary [HFDD])
Description: The HFDD items assess the number of mild, moderate, and severe HF experienced during the day and during the night. Mild HF are defined as a "sensation of heat without sweating", moderate HF are defined as a "sensation of heat with sweating, but able to continue activity", and severe HF are defined as a "sensation of heat with sweating, causing cessation (stopping) of activity".
Time Frame: Baseline to Week 12
Population: All randomized participants with data available at the time of evaluation.
Measure: Mean (Standard Deviation); unit: Number of HF
Arm/Group | Elinzanetant (BAY3427080) | Placebo
Number analyzed (Participants) | 312 | 315
Number of HF
  Baseline | 6.71 (7.15) | 6.81 (6.15)
  Change from Baseline: number analyzed (Participants) | 258 | 278
  Change from Baseline | -5.40 (7.29) | -3.50 (4.96)
Statistical Analysis 1: Comparison: Elinzanetant (BAY3427080) vs Placebo; For category "Change from baseline"; Test type: Superiority; p < 0.0001, Mixed model repeated measures (MMRM) — The type I error rate was controlled at a one-sided α=0.025 level; Difference in LS-means = -1.55, 95% CI 2-sided [-2.04 to -1.05]

2. Secondary Outcome: Mean Change in Patient-reported Outcomes Measurement Information System Sleep Disturbance Short Form 8b (PROMIS SD SF 8b) Total T-score From Baseline Over Time.
Description: The PROMIS SD SF 8b includes 8 items assessing sleep disturbance over the past 7 days. Items assess sleep quality, sleep depth and restoration associated with sleep, perceived difficulties with getting to sleep or staying asleep and perceptions of the adequacy of and satisfaction with sleep. Participants respond to the items on a 5-point scale from "not at all", "never" or "very poor" to "very much", "always" or "very good". Four of the items are scored reversely. Individual item scores are aggregated to total raw scores which range from 8 to 40. Total raw scores are converted into T-scores for comparison with population norms, with a mean of 50 and standard deviation of 10. T-scores range from 28.9 to 76.5. For both raw and T-scores higher scores indicate greater severity of sleep disturbance. According to available score cut points from PROMIS developers, T-scores can be interpreted as indicating mild (55-59), moderate (60-69), or severe (>70) sleep disturbance.
Time Frame: Baseline to Week 56
Population: All randomized participants with data available at the time of evaluation.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Elinzanetant (BAY3427080) | Placebo
Number analyzed (Participants) | 270 | 274
T-score
  Baseline | 57.35 (6.66) | 57.96 (7.63)
  Change from baseline to Week 1: number analyzed (Participants) | 265 | 270
  Change from baseline to Week 1 | -5.19 (7.17) | -1.60 (5.39)
  Change from baseline to Week 2: number analyzed (Participants) | 262 | 265
  Change from baseline to Week 2 | -6.78 (7.96) | -2.89 (6.78)
  Change from baseline to Week 3: number analyzed (Participants) | 258 | 265
  Change from baseline to Week 3 | -7.67 (8.24) | -3.34 (6.88)
  Change from baseline to Week 4: number analyzed (Participants) | 249 | 263
  Change from baseline to Week 4 | -7.70 (8.27) | -3.81 (6.98)
  Change from baseline to Week 8: number analyzed (Participants) | 241 | 253
  Change from baseline to Week 8 | -7.98 (8.58) | -4.36 (7.64)
  Change from baseline to Week 12: number analyzed (Participants) | 228 | 246
  Change from baseline to Week 12 | -7.97 (8.04) | -5.26 (8.02)
  Change from baseline to Week 18: number analyzed (Participants) | 188 | 192
  Change from baseline to Week 18 | -8.83 (9.05) | -5.77 (7.82)
  Change from baseline to Week 24: number analyzed (Participants) | 178 | 195
  Change from baseline to Week 24 | -9.77 (9.00) | -5.85 (7.79)
  Change from baseline to Week 36: number analyzed (Participants) | 186 | 190
  Change from baseline to Week 36 | -9.20 (8.74) | -5.88 (8.38)
  Change from baseline to Week 52: number analyzed (Participants) | 151 | 159
  Change from baseline to Week 52 | -9.36 (8.41) | -5.73 (7.91)
  Change from baseline to Week 56 (Follow-up): number analyzed (Participants) | 184 | 177
  Change from baseline to Week 56 (Follow-up) | -5.83 (8.71) | -5.38 (7.50)

3. Secondary Outcome: Mean Change in Menopause Specific Quality of Life Scale (MENQOL) Total Score From Baseline Over Time
Description: The MENQOL questionnaire is comprised of 29 items assessing the presence of menopausal symptoms and the impact of menopause on health-related quality of life over the past week. The items assess four domains of symptoms and functioning: Vasomotor functioning, psychosocial functioning, physical functioning, and sexual functioning. For each item, the participant indicates if they have experienced the symptom (yes/no). If they select yes, they rate how bothered they were by the symptom using a six-point verbal descriptor scale, with response options ranging from 0 'not at all bothered' to 6 'extremely bothered'. Based on the individual responses, item scores, domain scores, and a total MENQOL score are calculated. Each score ranges from 1-8, higher scores indicate greater bother.
Time Frame: Baseline to Week 56
Population: All randomized participants with data available at the time of evaluation.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Elinzanetant (BAY3427080) | Placebo
Number analyzed (Participants) | 262 | 264
Scores on a scale
  Baseline | 4.10 (1.21) | 4.41 (1.37)
  Change from baseline to Week 4: number analyzed (Participants) | 235 | 250
  Change from baseline to Week 4 | -0.94 (1.22) | -0.67 (1.21)
  Change from baseline to Week 8: number analyzed (Participants) | 233 | 243
  Change from baseline to Week 8 | -1.07 (1.24) | -0.86 (1.18)
  Change from baseline to Week 12: number analyzed (Participants) | 220 | 235
  Change from baseline to Week 12 | -1.10 (1.25) | -0.95 (1.32)
  Change from baseline to Week 18: number analyzed (Participants) | 183 | 185
  Change from baseline to Week 18 | -1.30 (1.32) | -1.11 (1.40)
  Change from baseline to Week 24: number analyzed (Participants) | 173 | 185
  Change from baseline to Week 24 | -1.25 (1.17) | -1.15 (1.37)
  Change from baseline to Week 36: number analyzed (Participants) | 179 | 182
  Change from baseline to Week 36 | -1.18 (1.21) | -1.02 (1.42)
  Change from baseline to Week 52: number analyzed (Participants) | 147 | 154
  Change from baseline to Week 52 | -1.30 (1.33) | -1.11 (1.35)
  Change from baseline to Week 56 (Follow-up): number analyzed (Participants) | 178 | 172
  Change from baseline to Week 56 (Follow-up) | -0.82 (1.25) | -1.04 (1.59)

ADVERSE EVENTS:
Time Frame: Adverse events tables: up to 14 days from the last drug intake, up to 54 weeks. All-cause mortality table: after signing informed consent up to the last contact per participant, up to 62 weeks.
Description: 1 participant who was assigned to the elinzanetant arm received no study drug and was excluded from the SAF. In addition, 1 participant who was assigned to the placebo arm received a kit containing elinzanetant at the Week 8 visit and is therefore assigned to the elinzanetant arm in the SAF. SAF: Elinzanetant=313, Placebo=314.
Arm/Group | Elinzanetant (BAY3427080) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/313 | 0/314
Serious Adverse Events (participants affected / at risk) | 13/313 | 6/314
Other Adverse Events (participants affected / at risk) | 85/313 | 73/314
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elinzanetant (BAY3427080) (N=313) | Placebo (N=314)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Fusobacterium infection (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Meningitis meningococcal (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Encephalitis toxic (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elinzanetant (BAY3427080) (N=313) | Placebo (N=314)
Fatigue (General disorders) | 21 (23) | 9 (9)
COVID-19 (Infections and infestations) | 22 (22) | 32 (32)
Nasopharyngitis (Infections and infestations) | 15 (16) | 21 (23)
Headache (Nervous system disorders) | 30 (51) | 22 (51)
Somnolence (Nervous system disorders) | 16 (18) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will submit material for public dissemination to the sponsor at least 60 days prior to submission. The PI agrees that all reasonable comments made by the sponsor will be incorporated into the publication. The sponsor can request that the publication be delayed for up to 6 months and for an exceptional additional delay, if proprietary information and/or Intellectual Property Rights and Know-How might otherwise be compromised or lost.

DOCUMENTS (2):
  • Study Protocol (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT05030584/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT05030584/SAP_001.pdf